CLINICAL TRIAL: NCT03380741
Title: Molecular Diagnostics Using a Novel Lab-on-a-chip and MRI for Detecting Cervical Cancer
Brief Title: Lab-on-a-chip Detection of Cervical Cancer Tumour Markers
Acronym: MODULAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); St. George's NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR4868
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical/vaginal cytology swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group1: Tumour present on histology and MRI following biopsy/LLETZ
  Interventions: Diagnostic Test: Tumour markers detection
- Group 2: Tumour absent on MRI following biopsy/LLETZ
  Interventions: Diagnostic Test: Tumour markers detection
- Group 3: Tumour recurrence present at the vaginal vault on MRI
  Interventions: Diagnostic Test: Tumour markers detection
- Group 4: Tumour recurrence absent at the vaginal vault on MRI
  Interventions: Diagnostic Test: Tumour markers detection
- Group 5: Normal cervix at colposcopy
  Interventions: Diagnostic Test: Tumour markers detection

INTERVENTIONS:
Diagnostic Test: Tumour markers detection — Lab on a chip detection of tumour markers measured from vaginal/cervical cytology swab

SUMMARY:
This study aims to establish whether tumour markers measured from cytological samples can improve cervical cancer detection both prior to treatment and after treatment during follow up.

All patients with presumed early cervical cancer referred to the Gynaecological Oncology Unit at The Royal Marsden Hospital and patients previously surgically treated for early cervical cancer with a suspected recurrence will be invited to participate.

Women attending the Colposcopy Unit at St George's Hospital, with a normal cervix will be invited to participate.

An endovaginal receiver coil has been designed and developed at the Institute of Cancer Research and Royal Marsden NHS Foundation Trust for use at high field strengths (3T).

A cytology swab, similar to a smear test, will be used to collect a sample of cells to evaluate the presence of tumour markers.

The presence of tumour markers will be measured by a lab-on-a-chip and polymerase chain reaction (PCR) testing system.

DETAILED DESCRIPTION:
Cervical cytology: This will be done prior to MRI at an out-patient visit or at the scan visit in all study subjects with cancer. IN those patients with a normal cervix at colposcopy, the sample will be taken as part of the colposcopy examination. The procedure will be identical to that used for cervical smear testing and involves the insertion of a speculum and taking a swab from the cervix and/ or vaginal vault for tumour marker assessment on lab-on-a-chip. Additionally, the sample will be examined conventionally to assess cytology.

MRI scan: For patients with primary disease, this will be done using an endovaginal technique. A ring design endovaginal coil will be inserted endovaginally around the cervix. It acts as a dedicated receiver, and the substantially improved signal enables high-spatial resolution images to be obtained (voxel size < 0.5 mm3). In patients being followed up after definitive surgery, in whom recurrence is suspected, MRI will be done using a standard phased array technique if the cervix is absent. In both instances, the MRI sequences will be standard and involve the use of T2-W and diffusion weighted sequences in 3 orthogonal planes. Contrast agents will not be administered. Intramuscular antiperistaltic agents (20 mg hyoscine butylbromide) are used routinely for pelvic imaging.

Histological analysis: Biopsies will be obtained from all patients with primary disease. This will be either a cone or LLETZ biopsy. In some cases with clearly visualized tumour due for radical hysterectomy, a punch biopsy may suffice for diagnosis.

In patients with suspected recurrence, a biopsy will be obtained if feasible and a visible mass is evident on imaging. In cases without a visible mass, or if biopsy is not feasible, vault cytology will be use as the gold standard. In the absence of adequate histology or cytology for validating the presence or absence of tumour, the patient will be withdrawn from the study.

Data Recording: Patient data will be recorded on case report forms. Patient data from case report forms will be recorded on a password protected study database. The MRI images will be placed onto the hospital picture archiving and communications system (PACS) and clinical reports will be available immediately to the referring clinicians.

Good Clinical Practice: The trial will be conducted in compliance with the protocol, standard operating procedures, policies, local R&D management guidance, Good Clinical Practice including the Research Governance Framework 2005 including the current Human Tissue Act, Human Tissue (Quality and Safety for Human Application) Regulations, the Medical Devices Regulations and Ionising Radiation (Medical Exposures) Regulations.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with presumed early stage cervical cancer (squamous or adenocarcinoma on histology) being considered for curative surgery.

  * Patients treated surgically for cervical cancer (squamous or adenocarcinoma on histology) being followed-up for suspected recurrent disease.
  * Patients with normal cervix at colposcopy examination.

Exclusion Criteria:

* Ferromagnetic metal implants, claustrophobia (MRI incompatibility). Neuroendocrine or unusual histological subtypes. Abnormal cervix seen at colposcopy examination (for Normal cervix cohort).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with presumed early cervical cancer referred to the Gynaecological Oncology Units at The Royal Marsden Hospital and patients previously surgically treated for early cervical cancer currently undergoing follow up with suspected cancer recurrence will be invited to participate.
  Women attending St George's Hospital colposcopy clinic, who are judged to have a normal cervix on colposcopy examination will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Lab-on-a-chip agreement with PCR system | 20 months
  To compare the agreement (sensitivity/specificity) between lab-on-a-chip system and PCR system in detecting tumour markers (HPV and cancer-specific gene overexpression) derived from patients with biopsy/cytology proven i) primary and ii) recurrent squamous or adeno cervical cancer and those from cytologically normal cervix.

SECONDARY OUTCOMES:
Primary disease | 20 months
  To determine the sensitivity of tumour markers (HPV and cancer-specific gene overexpression) derived from lab-on-a-chip system in patients with primary cervical cancer (versus histology as the gold standard).
Recurrent disease | 20 months
  To determine the sensitivity of tumour markers (HPV and cancer-specific gene overexpression) derived from lab-on-a-chip system in patients with recurrent cervical cancer (versus histology as the gold standard).
Exploratory radiomic outcome | 20 months
  To determine association/correlation between radiomic features of tumour identified on endovaginal MRI with tumour markers (HPV and cancer-specific gene overexpression).

IPD SHARING:
Plan to Share IPD: No